CLINICAL TRIAL: NCT04854239
Title: Accuracy of Half-guided Implant Placement With Machine-driven or Manual Insertion: a Prospective, Randomized Clinical Study
Brief Title: Accuracy of Half-guided Implant Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: NSK Europe GmbH (Industry); Botiss Medical AG (Other); Institut Straumann AG (Industry); Dicomlab Kft. (Unknown); Hungarian Human Resources Development Operational Program (EFOP-3.6.2-16-2017-00006) (Unknown); Excellence Program of the Ministry for Innovation and Technology in Hungary (Unknown)
Responsible Party: Principal Investigator, Balint Molnar, Dr. Balint Molnar DMD, PhD, associate professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Accuracy-Semmelweis-Perio
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Partial-edentulism
Keywords: dental implants; computer-assisted surgery; guided surgery; accuracy; machine driven implant insertion; manual implant insertion

STUDY DESIGN:
Intervention Model Description: Forty patients were treated; implant insertion with half-guided surgical protocol was utilized by surgical motor (20 patients, machine-driven group) or torque wrench (20 patients, manual group) in the maxilla.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were not aware whether implant were placed with a contra-angled handpiece or with a torque wrench. 3D implant position accuracy evaluation was performed blinded, randomization sequence was revealed after analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Machine-driven group (Experimental): In the machine-driven group, after guided implant bed preparation, implant insertion was performed with contra-angled handpiece.
  Interventions: Procedure: Half-guided implant placement
- Manual group (Experimental): In the manual group, after guided implant bed preparation, implant insertion was performed with torque-wrench.
  Interventions: Procedure: Half-guided implant placement

INTERVENTIONS:
Procedure: Half-guided implant placement — The surgery was performed under local anaesthesia in both groups, half-guided implant placement was carried out based on randomization.
  Other Names: Guided implant placement

SUMMARY:
The aim of the present prospective randomized controlled study is to compare the accuracy of implant placement performed either with a surgical motor or a torque wrench as part of a half-guided surgical protocol after maxillary sinus floor augmentation.

DETAILED DESCRIPTION:
Implant insertion with half-guided surgical protocol was utilized by surgical motor (machine-driven group) or torque wrench (manual group) in the maxilla. Forty patients were randomly divided in two study groups; 20 implants were inserted with a surgical motor and 20 implants with a torque wrench. After the healing period, accuracy comparison method between planned and actual implant positions was performed based on digital intraoral scan. Coronal, apical and angular deviation parameters, insertion time and maximum insertion torque was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* at least one edentulous maxillary premolar or molar site treated successfully by sinus floor elevation with a xenogenic bone substitute (cerabone, botiss biomaterials, Zossen, Germany) confirmed by preoperative cone-beam computed tomography
* full- mouth plaque and bleeding scores (FMPS and FMBS) <20%
* good patient compliance (including willingness to participate in the follow-up procedures)
* signed informed consent

Exclusion Criteria:

* clinically relevant diseases (e.g.: diabetes, rheumatism, cancer)
* systemic steroid or bisphosphonate use
* acute or chronic inflammatory processes

Ages: 29 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Global coronal implant position deviation | 3 months after implant placement
  Measurement: comparison of planned and actual implant position in a virtual model. Tool: Linear measurement with Amira 5.4.0 (Thermo Fisher Scientific, USA). Unit: mm
Global apical implant position deviation | 3 months after implant placement
  Measurement: comparison of planned and actual implant position in a virtual model. Tool: Linear measurement with Amira 5.4.0 (Thermo Fisher Scientific, USA). Unit: mm
Horizontal coronal implant position deviation | 3 months after implant placement
  Measurement: comparison of planned and actual implant position in a virtual model. Tool: Linear measurement with Amira 5.4.0 (Thermo Fisher Scientific, USA). Unit: mm
Horizontal apical implant position deviation | 3 months after implant placement
  Measurement: comparison of planned and actual implant position in a virtual model. Tool: Linear measurement with Amira 5.4.0 (Thermo Fisher Scientific, USA). Unit: mm
Angular implant position deviation | 3 months after implant placement
  Measurement: comparison of planned and actual implant position in a virtual model. Tool: Linear measurement with Amira 5.4.0 (Thermo Fisher Scientific, USA). Unit: mm

SECONDARY OUTCOMES:
Implant insertion torque | During implant insertion
  Measurement: Insertion torque. Tool: torque wrech Unit: Ncm
Implant insertion torque | During implant insertion
  Measurement: Insertion torque. Tool: surgical motor Unit: Ncm
Duration of implant insertion | During implant insertion
  Measurement: Duration of implant insertion Tool: stopwatch Unit: seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orban K, Varga E Jr, Windisch P, Braunitzer G, Molnar B. Accuracy of half-guided implant placement with machine-driven or manual insertion: a prospective, randomized clinical study. Clin Oral Investig. 2022 Jan;26(1):1035-1043. doi: 10.1007/s00784-021-04087-0. Epub 2021 Aug 16. PMID 34401946